CLINICAL TRIAL: NCT03230838
Title: A Phase 2, Randomized, Active Comparator-Controlled, Multicenter, Double-Blind Clinical Trial to Study the Safety and Efficacy of Ceftolozane/Tazobactam (MK-7625A) Versus Meropenem in Pediatric Subjects With Complicated Urinary Tract Infection, Including Pyelonephritis
Brief Title: MK-7625A Versus Meropenem in Pediatric Participants With Complicated Urinary Tract Infection (cUTI) (MK-7625A-034)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 7625A-034; 2016-004153-32 (EudraCT Number)
Record Dates: First submitted 2017-07-24; First posted 2017-07-26 (Actual); Results first posted 2021-12-01 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-05

CONDITIONS: Complicated Urinary Tract Infection; Pyelonephritis
MeSH Terms: conditions — Pyelonephritis | interventions — ceftolozane, tazobactam drug combination; Meropenem

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Ceftolozane/Tazobactam (Experimental): Ceftolozane 20 mg/kg and tazobactam 10 mg/kg (maximum 1 g and 0.5 g/dose) administered intravenously (IV) every 8 hours for 7-14 days
  Interventions: Drug: Ceftolozane/Tazobactam
- Meropenem (Active Comparator): Meropenem 20 mg/kg (maximum 1 g/dose) administered IV every 8 hours for 7-14 days
  Interventions: Drug: Meropenem

INTERVENTIONS:
Drug: Ceftolozane/Tazobactam — 12 to <18 years of age: Ceftolozane 1 g/dose; Tazobactam 0.5 g/dose via a 60-minute (±10 minutes) IV infusion every 8 hours for 7-14 days. <12 years of age: Ceftolozane 20 mg/kg with Tazobactam 10 mg/kg (not to exceed Ceftolozane 1 g and Tazobactam 0.5 g) via a 60-minute (±10 minutes) IV infusion every 8 hours for 7-14 days.
  Arms: Ceftolozane/Tazobactam
Drug: Meropenem — Meropenem 20 mg/kg (maximum 1 g/dose) administered IV every 8 hours for between 7 to 14 days.
  Other Names: MERREM®
  Arms: Meropenem

SUMMARY:
This study aims to evaluate the safety and tolerability of MK-7625A (ceftolozane/tazobactam) compared with that of meropenem in pediatric participants with cUTI, including pyelonephritis.

ELIGIBILITY:
Inclusion Criteria:

* Has a legally acceptable representative who provides documented informed consent / assent for the trial.
* Ages from birth (defined as >32 weeks gestational age and ≥7 days postnatal) to <18 years of age.
* Requires IV antibacterial therapy for the treatment of cUTI.
* Have a pretreatment baseline urine culture specimen obtained within 48 hours before the start of administration of the first dose of study treatment and preferably prior to administration of any potentially therapeutic antibiotics.
* Has pyuria.
* Has clinical signs and/or symptoms of cUTI at the Screening Visit.
* Is not of reproductive potential; but if of reproductive potential agrees to avoid becoming pregnant or impregnating a partner during screening, while receiving study treatment and for at least 30 days after the last dose of study treatment.
* Female of reproductive potential is not pregnant, and not planning to become pregnant within 30 days of the last day of treatment administration; and is nonlactating.

Exclusion Criteria:

* Is currently participating in or has participated in an interventional clinical trial with an investigational compound or device within 30 days prior to the first dose of study treatment in this current trial.
* Has previously participated in any trial of ceftolozane or ceftolozane/tazobactam or has enrolled previously in the current trial and been discontinued.
* Has a history of any moderate or severe hypersensitivity (e.g.anaphylaxis), allergic reaction, or other contraindication to any of the following: β-lactam antibiotics (e.g, penicillins, cephalosporins, and carbapenems), β-lactamase inhibitors (e.g. tazobactam, sulbactam, clavulanic acid, avibactam), or metronidazole.
* Has a history of a cUTI within the past 1 year prior to randomization known to be caused by a pathogen resistant to either IV study treatment.
* Has a concomitant infection at the time of randomization that requires nonstudy systemic antibacterial therapy in addition to IV study treatment or oral step -down therapy.
* Has received potentially therapeutic antibacterial therapy for a duration more than 24 hours during the 48 hours preceding the first dose of study treatment.
* Has any of the following: a) intractable UTI or pyelonephritis infection at baseline that the Investigator anticipates would require more than 14 days of study treatment; b) confirmed fungal urinary tract infection at time of randomization; c) permanent indwelling bladder catheter or instrumentation including nephrostomy; d) current urinary catheter that is not scheduled to be removed before the end of all study treatment; e) complete, permanent obstruction of the urinary tract; f) suspected or confirmed perinephric or intrarenal abscess; g) documented ileal loop reflux; h) suspected or confirmed prostatitis, urethritis, or epididymitis; i) trauma to pelvis/urinary tract.
* Has moderate or severe impairment of renal function.
* Has a seizure disorder or is anticipated to be treated with divalproex sodium or valproic acid during the course of study treatment.
* Is receiving, or is expected to receive, any prohibited medications.
* Has any rapidly progressing disease or immediately life-threatening illness, including acute hepatic failure, respiratory failure, or septic shock.
* Has an immunocompromising condition.
* Has a history of malignancy ≤5 years prior to signing informed consent.
* Is planning to receive suppressive/prophylactic antibiotics with gram-negative activity after completion of study treatment.

Ages: 7 Days to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 134 (Actual)
Dates: Start 2018-04-26 (Actual); Primary Completion 2020-12-03 (Actual); Study Completion 2020-12-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (52):
- United States (9):
  - Children's Hospital - Los Angeles ( Site 2509), Los Angeles, California
  - Children's Hospital of Orange County ( Site 2502), Orange, California
  - Rady Children's Hospital-San Diego ( Site 2505), San Diego, California
  - Ann & Robert H. Lurie Children's Hospital of Chicago ( Site 2519), Chicago, Illinois
  - Our Lady of the Lake Hospital ( Site 2512), Baton Rouge, Louisiana
  - St. Louis Children's Hospital ( Site 2508), St Louis, Missouri
  - SUNY Upstate Medical University Hospital ( Site 2510), Syracuse, New York
  - Wake Forest Baptist Health ( Site 2520), Winston-Salem, North Carolina
  - Baylor College Of Medicine ( Site 2515), Houston, Texas
- Greece (5):
  - Pan and Aglaia Kyriakou Children s Hospital ( Site 0780), Athens, Attica
  - University of Athens - Aghia Sophia Childrens Hospital ( Site 0730), Athens, Attica
  - Athens University Hospital ATTIKON ( Site 0790), Athens, Attica
  - Hippokration General Hospital of Thessaloniki ( Site 0700), Thessaloniki, Thessaloníki
  - General University Hospital of Larissa ( Site 0740), Larissa, Thessaly
- Hungary (6):
  - PTE AOK Klinikai Kozpont ( Site 0809), Pécs, Baranya
  - SZTE Szent-Gyorgyi Albert Klinikai Kozpont ( Site 0804), Szeged, Csongrád megye
  - SzSzBMK es Egyetemi Oktatokorhaz Josa Andras Oktatokorhaz ( Site 0808), Nyíregyháza, Szabolcs-Szatmár-Bereg
  - Semmelweis Egyetem ( Site 0810), Budapest
  - Heim Pal Orszagos Gyermekgyogyaszati Intezet ( Site 0801), Budapest
  - Debreceni Egyetem Klinikai Kozpont ( Site 0803), Debrecen
- Mexico (4):
  - Hospital Civil de Guadalajara Fray Antonio Alcalde ( Site 1202), Guadalajara, Jalisco
  - Instituto Tecnologico y de Estudios Superiores de Monterrey ( Site 1204), Monterrey, Nuevo León
  - Instituto Nacional de Pediatria ( Site 1201), Mexico City
  - Hospital Infantil de Mexico Federico Gomez ( Site 1203), Mexico City
- Poland (6):
  - Wojewodzki Szpital Obserwacyjno Zakazny ( Site 1606), Bydgoszcz, Kuyavian-Pomeranian Voivodeship
  - Szpital Uniwersytecki nr 1 im. Dr. Antoniego Jurasza w Bydgoszczy ( Site 1600), Bydgoszcz, Kuyavian-Pomeranian Voivodeship
  - Wojewodzki Szpital Zespolony im. Rydgiera ( Site 1607), Torun, Kuyavian-Pomeranian Voivodeship
  - Uniw. Szpital Dzieciecy w Krakowie ( Site 1609), Krakow, Lesser Poland Voivodeship
  - SPZOZ im. Dzieci Warszawy w Dziekanowie Lesnym ( Site 1608), Łomianki, Masovian Voivodeship
  - Instytut Centrum Zdrowia Matki Polki ( Site 1602), Lodz, Łódź Voivodeship
- Romania (4):
  - Spitalul Clinic de Urgenta pentru Copii Maria Sklodowska Curie ( Site 1707), Bucharest, București
  - Spit. Cl. de Urg. Copii Cluj Napoca ( Site 1708), Cluj-Napoca, Cluj
  - Spitalul Clinic de Urgenta pentru Copii Brasov ( Site 1703), Brasov
  - Institutul National de Boli Infectioase Prof. Dr. Matei Bals ( Site 1706), Bucharest
- Russia (4):
  - Russian Pediatric Clinical Hospital ( Site 1808), Moscow, Moscow
  - St.Petersburg State Pediatric Medical University ( Site 1811), Saint Petersburg, Sankt-Peterburg
  - Smolensk Regional Clinical Hospital ( Site 1800), Smolensk, Smolensk Oblast
  - Regional Childrens Clinical Hospital ( Site 1805), Stavropol, Stavropol Kray
- South Africa (3):
  - Molotlegi Street ( Site 1903), Pretoria, Gauteng
  - Inkosi Albert Luthuli Central Hospital ( Site 1902), Durban, KwaZulu-Natal
  - Red Cross War Memorial Children's Hospital ( Site 1900), Cape Town, Western Cape
- Turkey (Türkiye) (4):
  - Cukurova Universitesi Tıp Fakultesi Balcalı Hastanesi ( Site 2200), Adana
  - Hacettepe Universitesi Tip Fakultesi Hastanesi ( Site 2201), Ankara
  - Eskisehir Osmangazi Unv. Tip Fakultesi ( Site 2202), Eskişehir
  - SBU Sariyer Hamidiye Etfal Egitim ve Arastirma Hastanesi ( Site 2203), Istanbul
- Ukraine (7):
  - SI Dnipropetrovsk Regional Children Clinical Hospital DOR ( Site 2402), Dnipro, Dnipropetrovsk Oblast
  - PI Kryvorizka city clinical hospital 8 ( Site 2408), Kryvyy Rig, Dnipropetrovsk Oblast
  - Ivano-Frankivsk Regional Children Clinical Hospital ( Site 2411), Ivano-Frankivsk, Ivano-Frankivsk Oblast
  - Reg. Clinical Center of Urology and Nephrology n.a. V. I. Shapoval ( Site 2410), Kharkiv, Kharkivs’ka Oblast’
  - Kharkiv City Children Hospital 16 ( Site 2414), Kharkiv, Kharkivs’ka Oblast’
  - National Children Specialised Hospital OHMADYT MOH Ukraine ( Site 2409), Kyiv, Kyivska Oblast
  - Municipal Institution City Children s Clinical Hospital of Poltava City Council ( Site 2404), Poltava, Poltava Oblast

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Roilides E, Ashouri N, Bradley JS, Johnson MG, Lonchar J, Su FH, Huntington JA, Popejoy MW, Bensaci M, De Anda C, Rhee EG, Bruno CJ. Safety and Efficacy of Ceftolozane/Tazobactam Versus Meropenem in Neonates and Children With Complicated Urinary Tract Infection, Including Pyelonephritis: A Phase 2, Randomized Clinical Trial. Pediatr Infect Dis J. 2023 Apr 1;42(4):292-298. doi: 10.1097/INF.0000000000003832. Epub 2023 Jan 23. PMID 36689671

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Males and females from birth (>32 weeks gestational age and ≥7 days postnatal), to <18 years of age with complicated urinary tract infection (cUTI), including pyelonephritis, were enrolled in this study.
Period: Overall Study
Arm/Group | Ceftolozane/Tazobactam | Meropenem
Started | 101 | 33
Treated | 100 | 33
Completed | 97 | 33
Not Completed | 4 | 0
Not completed — Withdrawal by Subject | 3 | 0
Not completed — Temperature excursion | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ceftolozane/Tazobactam | Meropenem | Total
Number analyzed (Participants) | 101 | 33 | 134
Age, Continuous [Mean (Standard Deviation); unit: Years] | 5.3 (5.3) | 5.5 (5.7) | 5.4 (5.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 65 | 20 | 85
  Male | 36 | 13 | 49
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9 | 5 | 14
  Not Hispanic or Latino | 81 | 27 | 108
  Unknown or Not Reported | 11 | 1 | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 100 | 33 | 133
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With ≥1 Adverse Events (AEs)
Description: An adverse event (AE) is any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a medicinal product or protocol specified procedure, whether or not considered related to the medicinal product or protocol specified procedure. Any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a preexisting condition that is temporally associated with the use of the Sponsor's product, is also an AE.
Time Frame: Up to Day 88
Population: All randomized participants who received any amount of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Ceftolozane/Tazobactam | Meropenem
Number analyzed (Participants) | 100 | 33
Participants | 59 | 20
Statistical Analysis 1: Comparison: Ceftolozane/Tazobactam vs Meropenem; Difference in Percentage (C/T minus Mero); Test type: Other — The Miettinen & Nurminen method was used; Percentage Difference = -1.6, 95% CI 2-sided [-19.7 to 17.9] — Ceftolozane/Tazobactam (C/T) minus Meropenem (Mero)

2. Primary Outcome: Number of Participants Discontinuing Study Therapy Due to AE
Description: as for outcome 1
Time Frame: Up to Day 15
Population: All randomized participants who received any amount of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Ceftolozane/Tazobactam | Meropenem
Number analyzed (Participants) | 100 | 33
Participants | 1 | 0
Statistical Analysis 1: Comparison: Ceftolozane/Tazobactam vs Meropenem; Difference in Percentage (C/T minus Mero); Test type: Other — The Miettinen & Nurminen method was used; Percentage Difference = 1.0, 95% CI 2-sided [-9.5 to 5.5] — C/T minus Mero

3. Secondary Outcome: Percentage of Participants With a Clinical Response of Cure at the Test of Cure Visit
Description: Clinical response of cure is complete resolution or marked improvement in signs and symptoms of the complicated urinary tract infection (cUTI) or return to pre-infection signs and symptoms, such that no further antibiotic therapy (IV or oral) is required for the treatment of the cUTI. The 95% confidence intervals (CIs) of each treatment are unstratified Wilson CIs.
Time Frame: Up to Test of Cure Visit (up to 35 days)
Population: All randomized participants who received any amount of study treatment and have at least 1 acceptable causative uropathogen identified from a study-qualifying baseline urine culture.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Ceftolozane/Tazobactam | Meropenem
Number analyzed (Participants) | 71 | 24
Percentage of participants | 88.7 [79.31 to 94.18] | 95.8 [79.76 to 99.26]
Statistical Analysis 1: Comparison: Ceftolozane/Tazobactam vs Meropenem; Difference in Percentage (C/T minus Mero); Test type: Other — The Miettinen & Nurminen method stratified by age group with Cochran- Mantel-Haenszel (CMH) weights was used. If there was a zero count in any class of the stratum, the groups with the lower count were pooled with its near age group stratum in the model; Percentage Difference = -7.3, 95% CI 2-sided [-17.99 to 10.05] — C/T minus Mero

4. Secondary Outcome: Percentage of Participants With a Clinical Response of Cure at the End of Treatment Visit
Description: Clinical response of cure is complete resolution or marked improvement in signs and symptoms of the cUTI or return to pre-infection signs and symptoms, such that no further antibiotic therapy (IV or oral) is required for the treatment of the cUTI. The 95% CIs of each treatment are unstratified Wilson CIs.
Time Frame: Up to 48 hours after last oral dose (up to 19 days)
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Ceftolozane/Tazobactam | Meropenem
Number analyzed (Participants) | 71 | 24
Percentage of participants | 94.4 [86.39 to 97.79] | 100.0 [86.20 to 100.00]
Statistical Analysis 1: Comparison: Ceftolozane/Tazobactam vs Meropenem; Difference in Percentage (C/T minus Mero); Test type: Other — [test comment as in outcome 3, analysis 1]; Percentage Difference = -5.6, 95% CI 2-sided [-14.09 to 8.88] — C/T minus Mero

5. Secondary Outcome: Percentage of Participants With Microbiological Eradication of All Baseline Pathogens at the Test of Cure Visit
Description: Microbiological eradication of all baseline pathogens is defined as a postbaseline urine culture shows all uropathogens found at baseline at ≥10^5 colony-forming units (CFU)/mL are reduced to <10^4 CFU/mL. The 95% CIs of each treatment are unstratified Wilson CIs.
Time Frame: Up to Test of Cure Visit (up to 35 days)
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Ceftolozane/Tazobactam | Meropenem
Number analyzed (Participants) | 71 | 24
Percentage of participants | 84.5 [74.35 to 91.12] | 87.5 [69.00 to 95.66]
Statistical Analysis 1: Comparison: Ceftolozane/Tazobactam vs Meropenem; Difference in Percentage (C/T minus Mero); Test type: Other — [test comment as in outcome 3, analysis 1]; Percentage Difference = -3.0, 95% CI 2-sided [-17.13 to 17.40] — C/T minus Mero

6. Secondary Outcome: Percentage of Participants With Microbiological Eradication of All Baseline Pathogens at the End of Treatment Visit
Description: as for outcome 5
Time Frame: Up to 48 hours after last oral dose (up to 19 days)
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Ceftolozane/Tazobactam | Meropenem
Number analyzed (Participants) | 71 | 24
Percentage of participants | 93.0 [84.55 to 96.95] | 95.8 [79.76 to 99.26]
Statistical Analysis 1: Comparison: Ceftolozane/Tazobactam vs Meropenem; Difference in Percentage (C/T minus Mero); Test type: Other — The Miettinen & Nurminen method stratified by age group with CMH weights was used. If there was a zero count in any class of the stratum, the groups with the lower count were pooled with its near age group stratum in the model; Percentage Difference = -3.4, 95% CI 2-sided [-12.67 to 13.41] — C/T minus Mero

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs): From treatment (Day 1) up to 88 days. All-cause mortality: From randomization (Day 1) up to 88 days.
Description: For all-cause mortality the population analyzed was all randomized participants. For AEs the population analyzed was all randomized participants who received any amount of study treatment.
Groups:
- Ceftolozane/Tazobactam: Ceftolozane 20 mg/kg and tazobactam 10 mg/kg (maximum 1 g and 0.5 g/dose) administered IV every 8 hours for 7-14 days.
Arm/Group | Ceftolozane/Tazobactam | Meropenem
All-Cause Mortality (participants affected / at risk) | 0/101 | 0/33
Serious Adverse Events (participants affected / at risk) | 3/100 | 2/33
Other Adverse Events (participants affected / at risk) | 25/100 | 10/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ceftolozane/Tazobactam (N=100) | Meropenem (N=33)
Pyrexia (General disorders) | 0 (0) | 1 (1)
Pyelonephritis (Infections and infestations) | 1 (1) | 0 (0)
Pyelonephritis acute (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ceftolozane/Tazobactam (N=100) | Meropenem (N=33)
Thrombocytosis (Blood and lymphatic system disorders) | 7 (7) | 3 (3)
Diarrhoea (Gastrointestinal disorders) | 7 (7) | 3 (3)
Pyrexia (General disorders) | 6 (9) | 0 (0)
Rhinitis (Infections and infestations) | 2 (2) | 2 (2)
Urinary tract infection (Infections and infestations) | 1 (1) | 3 (3)
Vulvovaginitis (Infections and infestations) | 0 (0) | 2 (2)
Alanine aminotransferase increased (Investigations) | 4 (4) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 4 (4) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts or presentations regarding this trial 45 days prior to submission for publication/presentation. Any information identified by the Sponsor as confidential must be deleted prior to submission; this confidentiality does not include efficacy and safety results.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-09-14): https://cdn.clinicaltrials.gov/large-docs/38/NCT03230838/Prot_SAP_000.pdf